CLINICAL TRIAL: NCT03828188
Title: A 12-week, Randomized, Double-blind, Placebo-controlled 2x2 Cross-over Design Human Trial to Evaluate the Efficacy and Safety of Red Ginseng Concentrated Powder on Improvement of Blood Triglyceride Level
Brief Title: Efficacy and Safety of Red Ginseng Concentrated Powder on Improvement of Blood Triglyceride Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: JAR-FHL-RG2
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Hyperlipidemias
Keywords: Red Ginseng Concentrated Powder; Hyperlipidemias; Clinical Trial
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Red Ginseng Concentrated Powder in 12 weeks → rest in 4 weeks → Placebo 12 weeks.
  * Red Ginseng Concentrated Powder: 2 times daily(4.9 g/day)
  * Placebo: Red Ginseng Concentrated Powder: 2 times daily(4.9 g/day)
  Interventions: Dietary Supplement: Red Ginseng Concentrated Powder; Dietary Supplement: Placebo
- group B (Experimental): Placebo 12 weeks→ rest in 4 weeks → Red Ginseng Concentrated Powder in 12 weeks.
  * Red Ginseng Concentrated Powder: 2 times daily(4.9 g/day)
  * Placebo: Red Ginseng Concentrated Powder: 2 times daily(4.9 g/day)
  Interventions: Dietary Supplement: Red Ginseng Concentrated Powder; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Red Ginseng Concentrated Powder — Red Ginseng Concentrated Powder(4.9 g/day) for 12 weeks.
Dietary Supplement: Placebo — Placebo for 12 weeks.

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Red Ginseng Concentrated Powder on Improvement of Blood Triglyceride Level.

DETAILED DESCRIPTION:
This study was a 12-week, randomized, double-blind, placebo-controlled 2x2 cross-over design human trial. 50 subjects which of 25 by group were randomly divided into Red Ginseng Concentrated Powder and a placebo group.(A total of 100 subjects completed the 2x2 cross-over study.)

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70 years with Triglyceride 120-200 mg/dL

Exclusion Criteria:

* Lipid lowering agent within past 6 months
* Those with clinically significant severe cardiovascular, endocrine, immune, respiratory, liver, biliary, renal and urinary tract, neuropsychiatry, musculoskeletal, inflammatory and hematologic and gastrointestinal disorders
* Persons with significant hypersensitivity reactions to ginseng and red ginseng
* Those with a history of gastrointestinal disorders (ex, Crohn's disease) or gastrointestinal surgery (excluding simple cecal surgery or hernia surgery) that may affect the absorption of a product for clinical trials
* Those who have received antipsychotic medication within 2 months before screening
* Those with a history of alcoholism or substance abuse
* Those who participated in other clinical trials within 2 months before screening
* Laboratory test by show the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Changes of Fasting triglyceride | 12 weeks
  Changes of Fasting triglyceride was assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Lipid metabolism indices | 30 weeks
  Lipid metabolism indices were assessed before and after the intervention. The lipid metabolism index should be measured by collecting blood while keeping fasting for 12 hours or more. The inspection items are as follows.
  * Total cholesterol, triglyceride, LDL-C, HDL-C, Non HDL-C, VLDL-C, free fatty acid, Apo A1, Apo B, hs-CRP
  * Non HDL-C and VLDL-C are calculated by the calculation formula, and the first digit of the decimal point is indicated.
  * Non HDL-C= Total cholesterol - HDL-C VLDL-C= Total cholesterol - (HDL-C + LDL-C)
Changes of Arteriosclerosis indices | 30 weeks
  It is calculated by the calculation formula using the lipid metabolism indicator test item. Round off the third decimal place to the second decimal place. The items are as follows:
  * Total cholesterol/HDL-C, LDL-C/HDL-C, triglycerid/HDL-C, (Total cholesterol - HDL-C)/HDL-C, Apo B/Apo A1
Changes of Carnitine (Serum) | 30 weeks
  Carnitine (Serum)[μmol/L] was assessed before and after the intervention.
Changes of lipoprotein lipase | 30 weeks
  lipoprotein lipase[ng/ml] was assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided